CLINICAL TRIAL: NCT03779711
Title: Phase IIb Study of Intramyocardial Injection of Autologous Umbilical Cord Blood Derived Mononuclear Cells During Stage II Surgical Repair of Right Ventricular Dependent Variants of Hypoplastic Left Heart Syndrome (AutoCell-S2)
Brief Title: Intramyocardial Injection of Autologous Umbilical Cord Blood Derived Mononuclear Cells During Surgical Repair of Hypoplastic Left Heart Syndrome
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Timothy J Nelson, MD, PhD (Other)
Collaborators: University of Oklahoma (Other); Children's Hospital of Philadelphia (Other); Children's Hospital Los Angeles (Other); Children's Hospital Colorado (Other); Children's Hospitals and Clinics of Minnesota (Other); Ochsner Health System (Other); Children's of Alabama (Other); Children's Hospital Medical Center, Cincinnati (Other)
Responsible Party: Sponsor-Investigator, Timothy J Nelson, MD, PhD, Program Director, ReGen Theranostics, Inc.
Organization: ReGen Theranostics, Inc. (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 18-004753
Record Dates: First submitted 2018-12-04; First posted 2018-12-19 (Actual); Results first posted 2025-07-08 (Actual); Last update posted 2025-07-08 (Actual); Status verified 2025-06

CONDITIONS: Hypoplastic Left Heart Syndrome
Keywords: Hypoplastic Left Heart Syndrome; HLHS; Congenital Heart Disease; Umbilical Cord Blood; UCB; Cord blood; Stem cells; Regenerative therapy; Stage II Glenn; Glenn Surgery; single ventricle
MeSH Terms: conditions — Hypoplastic Left Heart Syndrome; Heart Defects, Congenital; Univentricular Heart

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Treatment (Experimental): Autologous (self) mononuclear cells derived from umbilical cord blood and that meet all release criteria are injected into the surface of the right heart muscle to achieve the target dose of 1-3 million cells per kilogram body weight . This is a one time treatment at the time of Stage II Glenn surgery .
  Interventions: Biological: Autologous (self) mononuclear cells derived from umbilical cord blood; Procedure: Stage II Surgical repair
- Control (Active Comparator): Clinical data will be collected before, during and after the Stage II surgical standard of care procedure. Requires additional imaging studies at 3 months that are not standard of care in addition to some blood tests that would be beyond standard of care. Information will be collected to document the clinical outcomes and will be compared with the information from the group receiving the investigational treatment used in this study.
  Interventions: Procedure: Stage II Surgical repair

INTERVENTIONS:
Biological: Autologous (self) mononuclear cells derived from umbilical cord blood — The investigational product will be delivered into the right myocardium via sub-epicardial injections of 0.1 mL per kg body weight to achieve the target dose of 1-3 million TNC per kg body weight.at the time of Stage II surgical repair.
  Arms: Treatment
Procedure: Stage II Surgical repair — This operation usually is performed about six months after Stage I surgery to divert half of the blood to the lungs when circulation through the lungs no longer needs as much pressure from the ventricle. The shunt to the pulmonary arteries is disconnected and the right pulmonary artery is connected directly to the superior vena cava, the vein that brings deoxygenated blood from the upper part of the body to the heart. This sends half of the deoxygenated blood directly to the lungs without going through the ventricle.

SUMMARY:
Researchers want to better understand what happens to the heart when the stem cells are injected directly into the muscle of the right side of the heart during the Stage II palliative surgery for single ventricle patients with hypoplastic left heart syndrome (HLHS) or HLHS variant. Researchers want to see if there are changes in the heart's structure/function following this stem cell-based therapy and compared to children that have not had cell-based therapy.

DETAILED DESCRIPTION:
This is a Phase IIb trial to determine if the delivery of the autologous UCB-MNC product into the myocardium of the right ventricle of the heart at the time of Stage II surgical repair will provide an improvement in cardiac function, reaching growth and developmental milestones, and quality of life, while also providing a reduction in the cumulative days of hospitalization following Stage II surgical repair. Long-term improvement in cardiac function, reaching growth and developmental milestones, reaching Stage III surgical repair pre-op work-up, prolonging time to cardiac transplantation or death, and improving quality of life will also be determined.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of HLHS or HLHS variant with single right ventricular dependent CHD having undergone Stage I surgical repair and undergoing Stage II surgical repair.
* Less than 13 months of age at time of Stage II surgical repair
* Previous participation in the UCB collection protocol with autologous UCB-MNC product that is acceptable for use (treatment arm only)

Exclusion Criteria:

* History of DMSO reaction (treatment arm only).
* Parent(s) and/or legal guardian(s) unwilling to have their child participate or unwilling to follow the study procedures.
* Severe chronic diseases at the discretion of the treating physician.
* Extensive extra-cardiac syndromic features.
* Known history of cancer.
* Any of the following complications of his/her congenital heart disease:

  1. Any condition requiring urgent, or unplanned interventional procedure within 15 days prior to Stage II surgical repair, unless complete and full cardiac recovery is documented by site investigator
  2. Severe pulmonary hypertension (reported in the medical record as >70% systemic pressure)
  3. Other clinical concerns as documented by a site investigator that would predict (more likely to happen than not to happen) a risk of severe complications or very poor outcome, not directly related to the stem cell product or its injection procedure, during or after Stage II surgical repair.

Max Age: 12 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 95 (Actual)
Dates: Start 2019-06-06 (Actual); Primary Completion 2022-05-22 (Actual); Study Completion 2026-02 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Frank Cetta, MD, Principal Investigator — Mayo Clinic; Harold M. Burkhart, M.D., Principal Investigator — Children's Hospital Oklahoma University Medical Center; Joseph W. Rossano, M.D., Principal Investigator — Children's Hospital of Philadelphia; David M. Overman, M.D., Principal Investigator — Children's Minnesota; Ram Kumar Subramanyan, M.D., Ph.D., Principal Investigator — Children's Hospital Los Angeles; James Jaggers, M.D., Principal Investigator — Children's Hospital Colorado; Benjamin Peeler, M.D., Principal Investigator — Ochsner Health System; Waldemar Carlo, M.D., Principal Investigator — University of Alabama at Birmingham; James Tweddell, M.D., Principal Investigator — Children's Hospital Medical Center, Cincinnati
Locations (8):
- United States (8):
  - Children's of Alabama, Birmingham, Alabama
  - Children's Hospital of Los Angeles, Los Angeles, California
  - Children's Hospital Colorado, Aurora, Colorado
  - Ocshner Medical Center, New Orleans, Louisiana
  - Children's Hospitals of Minnesota, Minneapolis, Minnesota
  - Cincinnati Children's Hospital and Medical Center, Cincinnati, Ohio
  - Oklahoma University Medical Center, Oklahoma City, Oklahoma
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Gallego-Navarro C, Jaggers J, Burkhart HM, Carlo WF, Morales DL, Qureshi MY, Rossano JW, Hagen CE, Seisler DK, Peral SC, Nelson TJ. Autologous umbilical cord blood mononuclear cell therapy for hypoplastic left heart syndrome: a nonrandomized control trial of the efficacy and safety of intramyocardial injections. Stem Cell Res Ther. 2025 May 1;16(1):215. doi: 10.1186/s13287-025-04316-3. PMID 40312733
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were recruited from May 2019 through January 2022 from the following eight sites: Children's Hospital Colorado, Children's Hospital Los Angeles, Children's Hospital of Alabama, Children's Hospital of Philadelphia, Children's Hospitals and Clinics of Minnesota - Minneapolis, Cincinnati Children's Hospital Medical Center, Ochsner Medical Center Jefferson, and Oklahoma University Medical Center.
Period: Overall Study
Arm/Group | Treatment | Control
Started | 50 | 45
Completed | 40 | 41
Not Completed | 10 | 4

BASELINE CHARACTERISTICS:
Population: All enrolled subjects.
Groups:
- Total: Total of all reporting groups
Arm/Group | Treatment | Control | Total
Number analyzed (Participants) | 50 | 45 | 95
Age, Continuous [Mean (Standard Deviation); unit: months] | 5.1 (1.5) | 5.8 (2.2) | 5.4 (1.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 20 | 31
  Male | 39 | 25 | 64
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 11 | 14
  Not Hispanic or Latino | 43 | 28 | 71
  Unknown or Not Reported | 4 | 6 | 10
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 3 | 1 | 4
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 3 | 3 | 6
  White | 36 | 29 | 65
  More than one race | 3 | 2 | 5
  Unknown or Not Reported | 5 | 10 | 15
Fractional Area Change (%) [Mean (Standard Deviation); unit: percentage of area] — Population: 2 treatment subjects did not have a baseline FAC measurement recorded, due to poor Echo image.
  percentage of area
    number analyzed (Participants) | 48 | 45 | 93
    (all) | 41.2 (6.4) | 41.3 (5.8) | 41.2 (6.1)
Troponin T (ng/mL) [Mean (Standard Deviation); unit: ng/mL] — Population: 8 treated and 4 control subjects did not have baseline Troponin, due to site error in collecting the values.
  ng/mL
    number analyzed (Participants) | 42 | 41 | 83
    (all) | 0.065 (0.185) | 0.037 (0.052) | 0.051 (0.136)

OUTCOME MEASURES:

1. Primary Outcome: Change in Right Ventricular Cardiac Function Measured by Apical Fractional Area Change (FAC)
Description: Right ventricular cardiac function as measured by echocardiogram that includes studies for apical fractional area change (FAC). Measured by percent.
Time Frame: baseline, 3 months post-Stage II surgery
Population: All enrolled subjects with both a baseline and 3-month Fractional Area Change value as assessed by Echocardiogram.
Measure: Least Squares Mean (95% Confidence Interval); unit: percentage of area
Arm/Group | Treatment | Control
Number analyzed (Participants) | 40 | 41
percentage of area | -2.2258 [-3.8988 to -0.5527] | -2.5116 [-4.1641 to -0.8590]
Statistical Analysis 1: Comparison: Treatment vs Control; Analysis of covariance (ANCOVA), adjusted for baseline FAC, is used to assess change in FAC from baseline to 3-months post-surgery; Test type: Superiority; p = 0.8095, ANCOVA; adjusted for baseline FAC

2. Primary Outcome: Change in Right Ventricular Cardiac Function Measured by Circumferential Strain.
Description: Right ventricular cardiac function as measured by echocardiogram that includes studies for circumferential strain. Measured by percent.
Time Frame: baseline, 3 months post-Stage II surgery
Population: All enrolled subjects with both baseline and 3-month circumferential strain values as assessed by echocardiogram.
Measure: Least Squares Mean (95% Confidence Interval); unit: percentage of area
Arm/Group | Treatment | Control
Number analyzed (Participants) | 30 | 35
percentage of area | 1.3412 [-0.3101 to 2.9925] | 0.1704 [-1.3582 to 1.6990]
Statistical Analysis 1: Comparison: Treatment vs Control; Analysis of covariance (ANCOVA), adjusted for baseline circumferential strain, is used to assess change in circumferential strain from baseline to 3-months post-surgery; Test type: Superiority; p = 0.3029, ANCOVA; Adjusted for baseline circumferential strain

3. Primary Outcome: Change in Right Ventricular Cardiac Function Measured by Longitudinal Strain.
Description: Right ventricular cardiac function as measured by echocardiogram that includes studies for longitudinal strain. Measured by percent.
Time Frame: baseline, 3 months post-Stage II surgery
Population: All enrolled subjects with both baseline and 3-month longitudinal strain values as assessed by echocardiogram.
Measure: Least Squares Mean (95% Confidence Interval); unit: percentage of area
Arm/Group | Treatment | Control
Number analyzed (Participants) | 39 | 39
percentage of area | 0.5394 [-.06073 to 1.6860] | -1.2407 [-2.3873 to -0.09402]
Statistical Analysis 1: Comparison: Treatment vs Control; Analysis of covariance (ANCOVA), adjusted for baseline longitudinal strain, is used to assess change in longitudinal strain from baseline to 3-months post-surgery; Test type: Superiority; p = 0.0323, ANCOVA; Adjusted for baseline longitudinal strain

4. Primary Outcome: Change in Right Ventricular Cardiac Function Measured by Apical Fractional Area Change (FAC)
Description: as for outcome 1
Time Frame: baseline, 12 months post-Stage II surgery
Population: All enrolled subjects with both baseline and 12-month fractional area changes values, as assessed by echocardiogram.
Measure: Least Squares Mean (95% Confidence Interval); unit: percentage of area
Arm/Group | Treatment | Control
Number analyzed (Participants) | 33 | 32
percentage of area | -3.8975 [-5.6808 to -2.1143] | -4.4310 [-6.2419 to -2.6201]
Statistical Analysis 1: Comparison: Treatment vs Control; Analysis of covariance (ANCOVA), adjusted for baseline FAC, is used to assess change in FAC from baseline to 12-months post-surgery; Test type: Superiority; p = 0.6765, ANCOVA; Adjusted for baseline FAC

5. Secondary Outcome: Change in Right Ventricular Cardiac Function Measured by Apical Fractional Area Change (FAC)
Description: as for outcome 1
Time Frame: baseline pre-op, hospital discharge from Stage II surgery (an average of 1-6 weeks)
Population: All enrolled subjects with both baseline and discharge fractional area change values, as assessed by echocardiogram.
Measure: Least Squares Mean (95% Confidence Interval); unit: percentage of area
Arm/Group | Treatment | Control
Number analyzed (Participants) | 46 | 43
percentage of area | -1.8109 [-3.6744 to 0.05259] | -3.0902 [-5.0176 to -1.1628]
Statistical Analysis 1: Comparison: Treatment vs Control; Analysis of covariance (ANCOVA), adjusted for baseline FAC, is used to assess change in FAC from baseline to discharge; Test type: Superiority; p = 0.3456, ANCOVA; Adjusted for baseline FAC

6. Secondary Outcome: Cumulative Days of Hospitalization
Description: Cumulative days of hospitalization per patient following discharge for the Stage II surgical repair.
Time Frame: 1-month post Stage II surgery
Population: All enrolled subjects.
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Treatment | Control
Number analyzed (Participants) | 50 | 45
days | 13.2 (9.6) | 13.3 (9.1)
Statistical Analysis 1: Comparison: Treatment vs Control; Kruskal-Wallis test comparing number of days in hospital post stage-II surgery; Test type: Superiority; p = 0.7760, Kruskal-Wallis

7. Secondary Outcome: Change in Weight
Description: Change in weight between baseline and 3-months post Stage II surgery. Weight as measured by scale provided as part of standard of care by subject's provider. Measured at home by subject's caregiver using the same scale for every home measurement of body weight. Caregivers will be instructed by the site to use the same scale for every home measurement of body weight. Scales will vary based on the institution's standard name/type used.
Time Frame: baseline, 3-months post Stage II surgery
Population: All enrolled subjects with weight values at both baseline and 3-months.
Measure: Mean (Standard Deviation); unit: kg
Arm/Group | Treatment | Control
Number analyzed (Participants) | 44 | 39
kg | 1.4 (1.3) | 1.3 (0.7)
Statistical Analysis 1: Comparison: Treatment vs Control; Kruskal-Wallis test for change in weight from baseline to 3-months post-surgery; Test type: Superiority; p = 0.9563, Kruskal-Wallis

8. Secondary Outcome: Change in Heart Rate
Description: Change in heart rate between baseline and 3-months post Stage II surgery. Heart rate as measured at home by subject's caregiver as standard of care per subject's provider. Caregivers will be instructed by the site staff on the best way to perform.
Time Frame: baseline, 3-months post Stage II surgery
Population: All enrolled subjects with heart rate values at both baseline and 3-months.
Measure: Mean (Standard Deviation); unit: beats per minute
Arm/Group | Treatment | Control
Number analyzed (Participants) | 43 | 38
beats per minute | 3.2 (14.5) | 4.6 (21.2)
Statistical Analysis 1: Comparison: Treatment vs Control; Kruskal-Wallis test for change in heart rate from baseline to 3-months post-surgery; Test type: Superiority; p = 0.9095, Kruskal-Wallis

9. Secondary Outcome: Change in Oxygen Saturation
Description: Change in oxygen saturation between baseline and 3-months post Stage II surgery. Oxygen saturation as measured at home by subject's caregiver using the pulse oximetry device provided as standard of care by subject's provider. Caregivers will be instructed by the site to use the same pulse oximetry device for every home measurement of oxygen saturation.
Time Frame: baseline, 3-months post Stage II surgery
Population: All enrolled subjects with oxygen saturation values at both baseline and 3-months.
Measure: Mean (Standard Deviation); unit: percentage of saturation
Arm/Group | Treatment | Control
Number analyzed (Participants) | 40 | 36
percentage of saturation | 4.9 (7.3) | 5.7 (6.6)
Statistical Analysis 1: Comparison: Treatment vs Control; Kruskal-Wallis test for change in oxygen saturation from baseline to 3-months post-surgery; Test type: Superiority; p = 0.6391, Kruskal-Wallis

10. Secondary Outcome: Change in Weight
Description: Weight as measured by scale provided as part of standard of care by subject's provider. Measured at home by subject's caregiver using the same scale for every home measurement of body weight. Caregivers will be instructed by the site to use the same scale for every home measurement of body weight. Scales will vary based on the institution's standard name/type used.
Time Frame: baseline, every 6 months post-Stage II surgery
Population: Enrolled subjects with weight values available at each 6-month follow-up visit.
Measure: Mean (Standard Deviation); unit: kg
Arm/Group | Treatment | Control
Number analyzed (Participants) | 50 | 45
kg
  Baseline | 6.1 (0.80) | 6.2 (1.20)
  6-months: number analyzed (Participants) | 49 | 38
  6-months | 8.1 (1.35) | 8.4 (1.27)
  12-months: number analyzed (Participants) | 40 | 36
  12-months | 9.7 (1.38) | 9.6 (1.30)
  18-months: number analyzed (Participants) | 42 | 36
  18-months | 11.0 (1.49) | 10.9 (1.64)
  24-months: number analyzed (Participants) | 39 | 31
  24-months | 12.0 (1.92) | 12.2 (1.82)

11. Secondary Outcome: Change in Arrhythmia and Heart Failure Medication
Description: Changes in arrhythmia and heart failure medications will be recorded by caregiver on the concomitant medication diary throughout the subject's participation in the study starting at the time of consent.
Time Frame: 3-months post-surgery
Population: All enrolled subjects.
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment | Control
Number analyzed (Participants) | 50 | 45
Participants
  ACE Inhibitor: Decrease | 1 | 0
  ACE Inhibitor: Increase | 13 | 14
  ACE Inhibitor: Not Prescribed | 31 | 24
  ACE Inhibitor: Same | 5 | 7
  Aldosterone receptor antagonis: Decrease | 0 | 0
  Aldosterone receptor antagonis: Increase | 5 | 4
  Aldosterone receptor antagonis: Not Prescribed | 45 | 41
  Aldosterone receptor antagonis: Same | 0 | 0
  Antiarrythmic Class IC: Decrease | 0 | 0
  Antiarrythmic Class IC: Increase | 0 | 1
  Antiarrythmic Class IC: Not Prescribed | 48 | 44
  Antiarrythmic Class IC: Same | 2 | 0
  Antiarrythmic Class III: Decrease | 0 | 0
  Antiarrythmic Class III: Increase | 0 | 0
  Antiarrythmic Class III: Not Prescribed | 46 | 45
  Antiarrythmic Class III: Same | 4 | 0
  B-blocker: Decrease | 0 | 0
  B-blocker: Increase | 2 | 1
  B-blocker: Not Prescribed | 46 | 41
  B-blocker: Same | 2 | 3
  Endotelin receptor antagonist: Decrease | 0 | 0
  Endotelin receptor antagonist: Increase | 0 | 0
  Endotelin receptor antagonist: Not Prescribed | 49 | 44
  Endotelin receptor antagonist: Same | 1 | 1
  Loop diuretic: Decrease | 1 | 0
  Loop diuretic: Increase | 25 | 20
  Loop diuretic: Not Prescribed | 21 | 20
  Loop diuretic: Same | 3 | 5
  Na+/K+ ATPase inhibitor: Decrease | 1 | 0
  Na+/K+ ATPase inhibitor: Increase | 10 | 4
  Na+/K+ ATPase inhibitor: Not Prescribed | 34 | 32
  Na+/K+ ATPase inhibitor: Same | 5 | 9
  PDE-3 inhibitor: Decrease | 0 | 0
  PDE-3 inhibitor: Increase | 1 | 0
  PDE-3 inhibitor: Not Prescribed | 49 | 45
  PDE-3 inhibitor: Same | 0 | 0
  PDE-5 inhibitor: Decrease | 0 | 3
  PDE-5 inhibitor: Increase | 10 | 10
  PDE-5 inhibitor: Not Prescribed | 39 | 28
  PDE-5 inhibitor: Same | 1 | 4
  Thiazide diuretic: Decrease | 0 | 0
  Thiazide diuretic: Increase | 5 | 3
  Thiazide diuretic: Not Prescribed | 45 | 42
  Thiazide diuretic: Same | 0 | 0

12. Secondary Outcome: Stage III Surgical Repair
Description: The number of research subjects eligible for Stage III surgical repair
Time Frame: Stage III surgery pre-op, approx. 4 years
Reporting Status: Not Posted, anticipated posting 2026-02

13. Secondary Outcome: Total Time Until Listed for Cardiac Transplantation
Description: The number of days between Stage II surgery and listed on cardiac transplantation list.
Time Frame: up to Stage III surgery pre-op, approx. 4 years
Reporting Status: Not Posted, anticipated posting 2026-02

14. Secondary Outcome: Change in Right Ventricular Cardiac Function Measured by Apical Fractional Area Change (FAC)
Description: as for outcome 1
Time Frame: baseline, Stage III surgery pre-op
Reporting Status: Not Posted, anticipated posting 2026-02

15. Secondary Outcome: Total Time Until Death
Description: The number of days between Stage II surgery and death occurrence
Time Frame: approx 4 years
Reporting Status: Not Posted, anticipated posting 2026-02

16. Secondary Outcome: Cumulative Days of Hospitalization
Description: Cumulative days of hospitalization per patient following discharge for the Stage II surgical repair.
Time Frame: 3-months post Stage II surgery
Population: All enrolled subjects.
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Treatment | Control
Number analyzed (Participants) | 50 | 45
days | 20.7 (26.0) | 15.6 (15.9)
Statistical Analysis 1: Comparison: Treatment vs Control; Kruskal-Wallis test comparing number of days in hospital post stage-II surgery; Test type: Superiority; p = 0.8782, Kruskal-Wallis

ADVERSE EVENTS:
Time Frame: 4 years
Description: Specific Adverse Event Terms will not be reported.
Arm/Group | Treatment | Control
All-Cause Mortality (participants affected / at risk) | 4/50 | 3/45
Serious Adverse Events (participants affected / at risk) | 38/50 | 27/45
Other Adverse Events (participants affected / at risk) | 48/50 | 45/45
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (N=50) | Control (N=45)
Abdominal Distension (Gastrointestinal disorders) | 1 (1) | 0 (0)
Acidosis (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 1 (1) | 0 (0)
Adult respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Agitation (Psychiatric disorders) | 0 (0) | 1 (1)
Arterial thromboembolism (Vascular disorders) | 0 (0) | 1 (1)
Atrioventricular block complete (Cardiac disorders) | 0 (0) | 1 (1)
Bacteremia (Infections and infestations) | 1 (1) | 1 (1)
Blood and lymphatic system disorders - Other Specify (Blood and lymphatic system disorders) | 1 (1) | 2 (2)
Bronchial infection (Infections and infestations) | 0 (0) | 2 (2)
Bronchopulmonary hemorrhage (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Cardiac arrest (Cardiac disorders) | 0 (0) | 2 (2)
Cardiac disorders - Other specify (Cardiac disorders) | 19 (28) | 7 (11)
Chylothorax (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 2 (2)
Chylous ascites (Gastrointestinal disorders) | 1 (1) | 0 (0)
Colonic perforation (Gastrointestinal disorders) | 1 (1) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Cyanosis (Cardiac disorders) | 2 (2) | 0 (0)
Death NOS (Gastrointestinal disorders) | 2 (2) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 4 (4) | 2 (2)
Depressed level of consciousness (Nervous system disorders) | 1 (1) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 1 (1) | 0 (0)
Ear and labyrinth disorders - Other specify (Ear and labyrinth disorders) | 0 (0) | 2 (2)
Edema face (General disorders) | 0 (0) | 1 (1)
Encephalopathy (Nervous system disorders) | 0 (0) | 1 (1)
Enterocolitis infectious (Infections and infestations) | 1 (1) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Fever (General disorders) | 1 (1) | 0 (0)
Flu like symptoms (General disorders) | 1 (1) | 0 (0)
Gastric hemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastritis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastroesophageal reflux disease (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastrointestinal disorders - Other specify (Gastrointestinal disorders) | 5 (9) | 3 (3)
General disorders - Other specify (General disorders) | 1 (1) | 0 (0)
Heart failure (Cardiac disorders) | 4 (4) | 0 (0)
Hypertension (Vascular disorders) | 0 (0) | 1 (1)
Hypoglycemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypotension (Vascular disorders) | 1 (1) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 9 (15) | 5 (5)
Infections and infestations - Other specify (Infections and infestations) | 2 (2) | 5 (5)
Injury, poisoning and procedural complications - Other specify (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Intracranial hemorrhage (Nervous system disorders) | 1 (2) | 1 (1)
Intraoperative cardiac injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Ischemia cerebrovascular (Nervous system disorders) | 1 (1) | 1 (1)
Laryngospasm (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Mediastinal infection (Infections and infestations) | 1 (1) | 0 (0)
Metabolism and nutrition disorders - Other specify (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Multi-organ failure (General disorders) | 2 (2) | 0 (0)
Muscle weakness left-sided (Nervous system disorders) | 1 (1) | 0 (0)
Nervous system disorders - Other specify (Nervous system disorders) | 1 (1) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 3 (3)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Recurrent laryngeal nerve palsy (Nervous system disorders) | 1 (1) | 0 (0)
Renal and urinary disorders - Other specify (Renal and urinary disorders) | 1 (1) | 1 (1)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 4 (5) | 3 (3)
Respiratory, thoracic and mediastinal disorders - Other specify (Respiratory, thoracic and mediastinal disorders) | 8 (14) | 9 (15)
Right ventricular dysfunction (Cardiac disorders) | 5 (5) | 1 (1)
Seizure (Nervous system disorders) | 3 (3) | 0 (0)
Sepsis (Infections and infestations) | 1 (3) | 1 (1)
Sinus bradycardia (Cardiac disorders) | 1 (1) | 0 (0)
Sinus tachycardia (Cardiac disorders) | 1 (1) | 0 (0)
Spasticity (Nervous system disorders) | 1 (1) | 0 (0)
Spinal cord compression (Nervous system disorders) | 1 (1) | 0 (0)
Supraventricular tachycardia (Cardiac disorders) | 1 (1) | 0 (0)
Surgical and medical procedures - Other specify (Surgical and medical procedures) | 4 (4) | 2 (5)
Thromboembolic event (Vascular disorders) | 4 (5) | 1 (1)
Tricuspid valve disease (Cardiac disorders) | 1 (1) | 1 (1)
Upper respiratory infection (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 2 (2)
Ventricular tachycardia (Cardiac disorders) | 2 (2) | 0 (0)
Vomiting (Gastrointestinal disorders) | 3 (3) | 0 (0)
Weight loss (Investigations) | 2 (2) | 0 (0)
Wound complication (Injury, poisoning and procedural complications) | 1 (2) | 0 (0)
Wound dehiscence (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Wound infection (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (N=50) | Control (N=45)
Anemia (Blood and lymphatic system disorders) | 9 (9) | 2 (2)
Blood and lymphatic system disorders - Other, specify (Blood and lymphatic system disorders) | 4 (4) | 8 (11)
Leukocytosis (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Atrial flutter (Cardiac disorders) | 1 (1) | 0 (0)
Atrioventricular block complete (Cardiac disorders) | 1 (1) | 0 (0)
Cardiac disorders - Other, specify (Cardiac disorders) | 16 (22) | 20 (35)
Cyanosis (Cardiac disorders) | 5 (5) | 2 (2)
Heart failure (Cardiac disorders) | 0 (0) | 1 (1)
Paroxysmal atrial tachycardia (Cardiac disorders) | 3 (7) | 0 (0)
Pericardial effusion (Cardiac disorders) | 2 (2) | 1 (1)
Right ventricular dysfunction (Cardiac disorders) | 1 (1) | 1 (1)
Sinus bradycardia (Cardiac disorders) | 3 (4) | 2 (2)
Sinus tachycardia (Cardiac disorders) | 7 (12) | 2 (5)
Supraventricular tachycardia (Cardiac disorders) | 3 (3) | 0 (0)
Tricuspid valve disease (Cardiac disorders) | 1 (1) | 0 (0)
Ventricular arrhythmia (Cardiac disorders) | 2 (2) | 0 (0)
Ventricular tachycardia (Cardiac disorders) | 2 (2) | 0 (0)
Congenital, familial and genetic disorders - Other, specify (Congenital, familial and genetic disorders) | 1 (1) | 0 (0)
Ear and labyrinth disorders - Other, specify (Ear and labyrinth disorders) | 3 (5) | 0 (0)
Middle ear inflammation (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Adrenal insufficiency (Endocrine disorders) | 2 (2) | 0 (0)
Endocrine disorders - Other, specify (Endocrine disorders) | 1 (1) | 0 (0)
Eye disorders - Other, specify (Eye disorders) | 2 (4) | 0 (0)
Periorbital edema (Eye disorders) | 2 (3) | 1 (1)
Abdominal distension (Gastrointestinal disorders) | 1 (1) | 0 (0)
Ascites (Gastrointestinal disorders) | 1 (1) | 0 (0)
Colitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 4 (4) | 3 (3)
Diarrhea (Gastrointestinal disorders) | 2 (2) | 3 (3)
Dysphagia (Gastrointestinal disorders) | 2 (2) | 1 (1)
Gastroesophageal reflux disease (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastrointestinal disorders - Other, specify (Gastrointestinal disorders) | 12 (22) | 10 (13)
Ileus (Gastrointestinal disorders) | 1 (1) | 0 (0)
Pancreatitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Rectal fissure (Gastrointestinal disorders) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 10 (12) | 13 (17)
Edema face (General disorders) | 2 (2) | 2 (2)
Edema limbs (General disorders) | 1 (1) | 1 (1)
Fatigue (General disorders) | 1 (1) | 1 (1)
Fever (General disorders) | 14 (26) | 17 (23)
General disorders and administration site conditions - Other, specify (General disorders) | 3 (4) | 3 (3)
Generalized edema (General disorders) | 4 (4) | 2 (2)
Localized edema (General disorders) | 1 (1) | 0 (0)
Malaise (General disorders) | 1 (1) | 0 (0)
Non-cardiac chest pain (General disorders) | 0 (0) | 1 (1)
Pain (General disorders) | 4 (4) | 6 (6)
Hepatobiliary disorders - Other, specify (Hepatobiliary disorders) | 4 (4) | 1 (1)
Portal hypertension (Hepatobiliary disorders) | 1 (1) | 0 (0)
Allergic reaction (Immune system disorders) | 1 (1) | 0 (0)
Immune system disorders - Other, specify (Immune system disorders) | 1 (2) | 0 (0)
Bacteremia (Infections and infestations) | 1 (1) | 0 (0)
Catheter related infection (Infections and infestations) | 0 (0) | 1 (1)
Conjunctivitis (Infections and infestations) | 0 (0) | 1 (1)
Infections and infestations - Other, specify (Infections and infestations) | 8 (10) | 9 (13)
Otitis media (Infections and infestations) | 6 (11) | 5 (6)
Pharyngitis (Infections and infestations) | 0 (0) | 1 (1)
Rash pustular (Infections and infestations) | 1 (1) | 0 (0)
Rhinitis infective (Infections and infestations) | 1 (1) | 0 (0)
Sepsis (Infections and infestations) | 1 (1) | 0 (0)
Sinusitis (Infections and infestations) | 1 (1) | 0 (0)
Skin infection (Infections and infestations) | 1 (1) | 0 (0)
Thrush (Infections and infestations) | 1 (1) | 1 (1)
Tracheitis (Infections and infestations) | 1 (1) | 0 (0)
Upper respiratory infection (Infections and infestations) | 7 (7) | 7 (11)
Urinary tract infection (Infections and infestations) | 2 (2) | 0 (0)
Bruising (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Fracture (Injury, poisoning and procedural complications) | 2 (3) | 1 (1)
Injury, poisoning and procedural complications - Other, specify (Injury, poisoning and procedural complications) | 2 (2) | 2 (2)
Intraoperative hemorrhage (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Postoperative hemorrhage (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Spinal fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Platelet count decreased (Investigations) | 0 (0) | 2 (2)
Thyroid stimulating hormone increased (Investigations) | 1 (1) | 0 (0)
Weight loss (Investigations) | 0 (0) | 3 (3)
White blood cell decreased (Investigations) | 0 (0) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 2 (2) | 3 (3)
Hyperkalemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypoalbuminemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypocalcemia (Metabolism and nutrition disorders) | 2 (3) | 4 (4)
Hypokalemia (Metabolism and nutrition disorders) | 7 (9) | 7 (7)
Hypomagnesemia (Metabolism and nutrition disorders) | 3 (3) | 0 (0)
Hyponatremia (Metabolism and nutrition disorders) | 6 (7) | 2 (2)
Hypophosphatemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Metabolism and nutrition disorders - Other, specify (Metabolism and nutrition disorders) | 4 (4) | 4 (4)
Muscle weakness lower limb (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Musculoskeletal and connective tissue disorder - Other, specify (Musculoskeletal and connective tissue disorders) | 2 (3) | 2 (2)
Encephalopathy (Nervous system disorders) | 1 (1) | 0 (0)
Hydrocephalus (Nervous system disorders) | 1 (1) | 0 (0)
Ischemia cerebrovascular (Nervous system disorders) | 1 (1) | 0 (0)
Movements involuntary (Nervous system disorders) | 3 (3) | 0 (0)
Nervous system disorders - Other, specify (Nervous system disorders) | 2 (2) | 3 (3)
Seizure (Nervous system disorders) | 1 (1) | 0 (0)
Spinal cord compression (Nervous system disorders) | 1 (1) | 0 (0)
Transient ischemic attacks (Nervous system disorders) | 1 (1) | 0 (0)
Tremor (Nervous system disorders) | 1 (1) | 0 (0)
Agitation (Psychiatric disorders) | 9 (9) | 5 (6)
Anxiety (Psychiatric disorders) | 1 (1) | 0 (0)
Delirium (Psychiatric disorders) | 2 (2) | 0 (0)
Irritability (Psychiatric disorders) | 3 (3) | 1 (1)
Psychiatric disorders - Other, specify (Psychiatric disorders) | 0 (0) | 1 (1)
Acute kidney injury (Renal and urinary disorders) | 1 (1) | 1 (2)
Renal and urinary disorders - Other, specify (Renal and urinary disorders) | 3 (3) | 1 (1)
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Aspiration (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 0 (0)
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 12 (12) | 6 (6)
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Chylothorax (Respiratory, thoracic and mediastinal disorders) | 5 (5) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 4 (10)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Hoarseness (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 10 (11) | 9 (10)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 3 (3)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 11 (12) | 7 (7)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 3 (3)
Pulmonary edema (Respiratory, thoracic and mediastinal disorders) | 10 (10) | 18 (18)
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 6 (6)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 2 (2)
Respiratory, thoracic and mediastinal disorders - Other, specify (Respiratory, thoracic and mediastinal disorders) | 27 (37) | 24 (47)
Rhinorrhea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Stridor (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 2 (2)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1)
Eczema (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Skin and subcutaneous tissue disorders - Other, specify (Skin and subcutaneous tissue disorders) | 2 (4) | 9 (13)
Surgical and medical procedures - Other, specify (Surgical and medical procedures) | 3 (4) | 6 (12)
Capillary leak syndrome (Vascular disorders) | 0 (0) | 1 (1)
Hypertension (Vascular disorders) | 14 (14) | 16 (17)
Hypotension (Vascular disorders) | 8 (11) | 1 (1)
Peripheral ischemia (Vascular disorders) | 1 (1) | 0 (0)
Thromboembolic event (Vascular disorders) | 5 (5) | 1 (1)
Vascular disorders - Other, specify (Vascular disorders) | 1 (2) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2024-03-20): https://cdn.clinicaltrials.gov/large-docs/11/NCT03779711/Prot_SAP_000.pdf